CLINICAL TRIAL: NCT03237858
Title: Multiple Cardiac Sensors for the Management of Heart Failure
Acronym: MANAGE-HF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 92125179
Record Dates: First submitted 2017-07-20; First posted 2017-08-03 (Actual); Results first posted 2024-03-27 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2023-11

CONDITIONS: Heart Failure, Congestive
Keywords: heart failure; diagnostics; heart sounds; CRT-D; ICD; remote monitoring
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- HeartLogic ON (Active Comparator): ICD and CRT-D devices with HeartLogic alerts turned ON
  Interventions: Device: HeartLogic ON
- HeartLogic OFF (Placebo Comparator): ICD and CRT-D devices with HeartLogic alerts turned OFF
  Interventions: Device: HeartLogic OFF

INTERVENTIONS:
Device: HeartLogic ON — Remote management of patients with CRT-D or ICD devices and the HeartLogic diagnostic feature turned OFF
  Arms: HeartLogic ON
Device: HeartLogic OFF — Remote management of patients with CRT-D or ICD devices and the HeartLogic diagnostic feature turned ON
  Arms: HeartLogic OFF

SUMMARY:
The MANAGE-HF study is a multi-center, global, prospective, open label, multi-phase trial intended to evaluate the clinical efficacy of the HeartLogic heart failure diagnostic feature.

DETAILED DESCRIPTION:
Phase I of the MANAGE-HF trial is not randomized, and is intended to evaluate the clinical integration of HeartLogic for managing patients with heart failure. There are no endpoints.

Phase II of the MANAGE-HF trial will assess the clinical effectiveness of remote monitoring of heart failure patients with implanted CRT-D or ICD cardiac devices that contain the diagnostic feature HeartLogic. This feature uses S1 and S3 heart sounds, night time heart rate, thoracic impedance, and respiration to alert clinicians when a patient's heart failure is worsening. The MANAGE-HF study will compare remote monitoring using HeartLogic alerts to drive heart failure care against patients with remote monitoring but without HeartLogic alerts.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is age 18 or above, or of legal age to give informed consent
2. Implanted with an cardiac resynchronization therapy defibrillator (CRT-D) or implantable cardioverter-defibrillator (ICD) device that has HeartLogic
3. Current symptomatic heart failure or New York Heart Association Class II or III at the time of enrollment
4. Remotely monitored by LATITUDE 5.0 (or future versions)
5. Willing and capable of participating in all study visits and complying with medication/treatment requirements associated with this clinical study at an approved clinical study center.
6. Meet at least one of the three following conditions:

   * At least one documented hospitalization with a primary diagnosis of worsening for heart failure during the 12 months prior to enrollment; or
   * Unscheduled outpatient visit with IV diuretic therapy for acute worsening of HF during 90 days prior to enrollment; or
   * N-terminal-pro brain natriuretic peptide (NT-proBNP) greater than 600 pg/mL or brain natriuretic peptide (BNP) greater than 150 pg/mL at any time during 90 days prior to enrollment

Exclusion Criteria:

1. The subject is unable to sign or refuses to sign the patient informed consent
2. Symptomatic heart failure at rest or New York Heart Association Class IV at the time of enrollment
3. The subject is implanted with unipolar right atrial or right ventricular leads
4. Subject has received or is scheduled to receive a heart transplant or ventricular assist device within the next 6 months
5. Subject is pregnant or planning to become pregnant during the study
6. Subject is enrolled in any other concurrent study (without prior written approval from Boston Scientific, excluding registries)
7. Glomerular filtration rate <25 mL/min who are non-responsive to diuretic therapy or are on chronic renal dialysis
8. Regularly scheduled intravenous heart failure therapy (for example inotropes or diuretics)
9. A life expectancy of less than 12 months per clinician discretion
10. APPLICABLE TO PHASE II ONLY: Subject enrolled in Phase I of MANAGE-HF
11. APPLICABLE TO PHASE II ONLY: Subject has been managed with HeartLogic Alerts ON at anytime within the past 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2017-08-30 (Actual); Primary Completion 2020-07-21 (Actual); Study Completion 2020-07-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Hernandez, MD, Principal Investigator — Duke University
Locations (30):
- United States (27):
  - Heart Center Research, LLC, Huntsville, Alabama
  - Cardiology Associates of Northeast Arkansas, Jonesboro, Arkansas
  - University of Southern California Hospital, Los Angeles, California
  - Cardiovascular Consultants, Oakland, California
  - Sharp Memorial Hospital, San Diego, California
  - University of California, San Francisco, San Francisco, California
  - University of Colorado, Aurora, Colorado
  - Emory University Hospital, Atlanta, Georgia
  - Parkview Hospital, Inc., Fort Wayne, Indiana
  - Community Health Network, Indianapolis, Indiana
  - Advanced Cardiovascular Specialists, Shreveport, Louisiana
  - Centra Care Heart and Vascular Center, Cold Spring, Minnesota
  - United Heart and Vascular, Saint Paul, Minnesota
  - Catholic Medical Center, Manchester, New Hampshire
  - Strong Memorial Hospital of the University of Rochester, Rochester, New York
  - Montefiore Medical Center, The Bronx, New York
  - Duke University Medical Center, Durham, North Carolina
  - Rex Hospital, Raleigh, North Carolina
  - Lindner Center for Research and Education at Christ Hosp, Cincinnati, Ohio
  - Bethesda North Hospital, Cincinnati, Ohio
  - PeaceHealth Sacred Heart Medical Center, Springfield, Oregon
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - Cardiology Consultants of Philadelphia, Yardley, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Stern Cardiovascular, Germantown, Tennessee
  - Southeast Texas Clinical Research Center, Beaumont, Texas
  - Sentara Norfolk General Hospital, Norfolk, Virginia
- France (2):
  - L'Hôpital privé du Confluent, Nantes
  - CHU Pontchaillou, Rennes
- Universitätsklinikum Würzburg AöR, Würzburg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hernandez AF, Albert NM, Allen LA, Ahmed R, Averina V, Boehmer JP, Cowie MR, Chien CV, Galvao M, Klein L, Kwan B, Lam CSP, Ruble SB, Stolen CM, Stein K; MANAGE-HF Study. Multiple cArdiac seNsors for mAnaGEment of Heart Failure (MANAGE-HF) - Phase I Evaluation of the Integration and Safety of the HeartLogic Multisensor Algorithm in Patients With Heart Failure. J Card Fail. 2022 Aug;28(8):1245-1254. doi: 10.1016/j.cardfail.2022.03.349. Epub 2022 Apr 21. PMID 35460884
- [Derived] Heggermont WA, Van Bockstal K. HeartlogicTM: ready for prime time? Expert Rev Med Devices. 2022 Feb;19(2):107-111. doi: 10.1080/17434440.2022.2038133. Epub 2022 Feb 12. No abstract available. PMID 35129007
- See also: Multiple cArdiac seNsors for mAnaGEment of Heart Failure (MANAGE-HF) - Phase I Evaluation of the Integration and Safety of the HeartLogic Multisensor Algorithm in Patients With Heart Failure — https://pubmed.ncbi.nlm.nih.gov/35460884/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Manage-HF Phase I began recruitment in August of 2017 and completed recruitment in May of 2019. Last Patient Last visit for Phase I occurred in July of 2020. MANAGE HF Phase I was determined to be sufficient by FDA on January 31, 2023, and phase II was not started.
Groups:
- MANAGE-HF Phase I: Two hundred subjects were enrolled in Phase I of MANAGE-HF. One hundred forty-four subjects were followed until the last patient enrolled completed his or her12-month visit.
  Thirty-seven subjects withdrew and 19 subjects died.
Period: Overall Study
Arm/Group | MANAGE-HF Phase I
Started | 200
Completed | 144
Not Completed | 56
Not completed — Death | 19
Not completed — Withdrawal by Subject | 37

BASELINE CHARACTERISTICS:
Population: There were 200 subjects enrolled and 191 completed the baseline visit. Demographics, medical history, physical assessment, heart failure assessment, and blood labs were taken at the baseline visit.
Arm/Group | MANAGE-HF Phase I
Number analyzed (Participants) | 191
Age, Continuous [Mean (Standard Deviation); unit: years] | 67 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62
  Male | 129
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 28
  White | 142
  More than one race | 0
  Unknown or Not Reported | 19
Region of Enrollment [Number; unit: participants]
  United States | 171
  France | 14
  Germany | 6
Heart Failure Hospitalization [Count of Participants; unit: Participants] | 112
Ischemic Heart Disease [Count of Participants; unit: Participants] | 90
Dilated Cardiomyopathy [Count of Participants; unit: Participants] | 75
Idiopathic Cardiomyopathy [Count of Participants; unit: Participants] | 20
Valvular disease [Count of Participants; unit: Participants] | 48
Valvular surgery [Count of Participants; unit: Participants] | 17
Thoracic surgery [Count of Participants; unit: Participants] | 18
Previous Myocardial Infarction [Count of Participants; unit: Participants] | 73
CABG [Count of Participants; unit: Participants] | 49
QRS duration (ms) [Mean (Standard Deviation); unit: ms] | 135 (31)
LVEF (%) [Mean (Standard Deviation); unit: %] | 25.6 (9.5)
RVEF (%) [Mean (Standard Deviation); unit: %] | 49.3 (12.5)
Chronic Obstructive Pulmonary Disease [Number; unit: participants] | 28
Asthma [Count of Participants; unit: Participants] | 12
Pulmonary hypertension [Count of Participants; unit: Participants] | 14
Pulmonary diseases other [Count of Participants; unit: Participants] | 13
Peripheral Vascular Disease [Count of Participants; unit: Participants] | 25
Renal dysfunction [Count of Participants; unit: Participants] | 50
Hypertension [Count of Participants; unit: Participants] | 144
Diabetes [Count of Participants; unit: Participants] | 69

OUTCOME MEASURES:

1. Primary Outcome: Manage-HF Phase I
Description: Phase-I was a single arm non-randomized study used to evaluate and optimize HeartLogic clinical integration and alert management. Phase-I had no outcome measures.
Time Frame: Data was collected from the time of consent until the last Phase I subject had completed their 12-month visit
Population: Manage-HF Phase II was not started, the trial was closed after phase I
Measure: Count of Participants; unit: Participants
Groups:
- MANAGE-HF Phase I: Number of participants contributing to the knowledge of the clinical integration of HeartLogic and the alert management process
Arm/Group | MANAGE-HF Phase I
Number analyzed (Participants) | 191
Participants | 191

ADVERSE EVENTS:
Time Frame: Adverse Events were collected for all enrolled subjects from the time of consent until the last Phase I subject had completed their 12-month visit
Description: Manage-HF Phase II was not started, the study was closed after Phase I
Groups:
- MANAGE-HF Phase I: MANAGE-HF Phase I was an open label, non-randomized single arm study
Arm/Group | MANAGE-HF Phase I
All-Cause Mortality (participants affected / at risk) | 19/200
Serious Adverse Events (participants affected / at risk) | 100/200
Other Adverse Events (participants affected / at risk) | 104/200
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MANAGE-HF Phase I (N=200)
Pulse Generator (Cardiac disorders) | 0 (0)
RA Lead (Cardiac disorders) | 0 (0)
RV Lead (Cardiac disorders) | 0 (0)
Cardiovascular-HF (Cardiac disorders) | 50 (92)
Cardiovascular-Non-HF (Cardiac disorders) | 55 (79)
Non-cardiovascular (Cardiac disorders) | 63 (130)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MANAGE-HF Phase I (N=200)
Pulse Generator (Cardiac disorders) | 0 (0)
RA Lead (Cardiac disorders) | 0 (0)
RV Lead (Cardiac disorders) | 0 (0)
Cardiovascular-HF (Cardiac disorders) | 82 (227)
Cardiovascular-Non-HF (Cardiac disorders) | 51 (83)
Non-cardiovascular (Cardiac disorders) | 30 (59)

LIMITATIONS AND CAVEATS:
Patients that were included in Phase I of MANAGE-HF were required to meet inclusion and exclusion criteria. This included evidence of worsened heart failure prior to enrollment, patients with severe kidney impairment or short life expectancy were excluded. Thus, the results are limited to the population that was studied. Furthermore, the small sample size and lack of a control group severely limits the interpretation of the results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-01): https://cdn.clinicaltrials.gov/large-docs/58/NCT03237858/Prot_SAP_000.pdf